CLINICAL TRIAL: NCT04825028
Title: Diagnostic Value of Angiography-derived Index of Microvascular Resistance in Coronary Artery Disease Patients and Its Prognostic Implication After Percutaneous Coronary Intervention
Brief Title: Diagnostic and Prognostic Value of Angiography-derived IMR
Acronym: CHART-MiCro
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Shanghai 10th People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZS-20210328
Record Dates: First submitted 2021-03-28; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Coronary Microvascular Dysfunction; Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Internal Diagnostic Accuracy Cohort: Consecutive patients with available CZT-SPECT within 3 months of measuring FFR in the left anterior descending coronary artery. In these patients, correlation between angiography-derived IMR and hyperemic microvascular resistance will be assessed.
  Interventions: Device: Angiography-drived Index of Microcirculatory Resistance
- External Diagnostic Accuracy Cohort: Patients are subgroup of previously published study (J Nucl Cardiol. 2020 Sep 30. doi: 10.1007/s12350-020-02252-8.), INOCA patients and normal controls confirmed by CZT-SPECT and angiography will be included for the assessment of angiography-derived IMR in diagnosing microvascular dysfunction.
  Interventions: Device: Angiography-drived Index of Microcirculatory Resistance
- Prognosis Cohort: Prognosis cohort, in which angiography-derived IMR will be measured in the target vessel after successful revascularization. Those patients have follow-up data after 2 years from index procedure.
  Interventions: Device: Angiography-drived Index of Microcirculatory Resistance

INTERVENTIONS:
Device: Angiography-drived Index of Microcirculatory Resistance — From coronary angiographic images, angiography-derived IMR will be calculated based on mathematical calculation.
  Angiography-derived IMR = (hyperemic Pa x angiography-derived FFR) x (vessel length / {K x V diastole}).
  Hyperemic Pa will be estimated from resting Pa according to prespecified equation.
  Other Names: Angio-IMR; CaIMR

SUMMARY:
The importance of the microvasculature in determining clinical outcomes has been highlighted in patients with coronary artery disease (CAD). For patients with stable CAD, despite the success of percutaneous coronary intervention (PCI) in relieving a stenosis in the epicardial coronary artery, microvascular dysfunction may preclude sufficient coronary flow and myocardial perfusion, possibly leading to worse clinical outcome. With the technical development of computational fluid dynamics, angiographic derivation of index of Index of Microcirculatory Resistance (IMR) without pressure wire, hyperemic agents, or theromdilution method is available as a potential alternative for pressure wire-derived IMR. In this regard, the current study will evaluate diagnostic implication of angiography-derived IMR and its prognostic implication after PCI in patients with stable CAD.

DETAILED DESCRIPTION:
The importance of the microvasculature in determining clinical outcomes has been highlighted in patients with coronary artery disease (CAD). For patients with stable CAD, despite the success of percutaneous coronary intervention (PCI) in relieving a stenosis in the epicardial coronary artery, microvascular dysfunction may preclude sufficient coronary flow and myocardial perfusion, possibly leading to worse clinical outcome. With the technical development of computational fluid dynamics, angiographic derivation of IMR without pressure wire, hyperemic agents, or theromdilution method is available as a potential alternative for pressure wire-derived IMR. In this regard, the current study will evaluate diagnostic implication of angiography-derived IMR and its prognostic implication after PCI in patients with stable CAD.

This study cohorts consist with 3 separate cohort: first, internal diagnostic accuracy cohort, which will evaluate correlation between angiography-derived IMR and hyperemic microvascular resistance calculated using Cadmium-Zinc-Telluride Single-Photon Emission Computed Tomography (CZT-SPECT)-derived myocardial blood flow and invasively measured pressure data. For this, 53 consecutive patients with available CZT-SPECT within 3 months of measuring FFR in the left anterior descending coronary artery will be evaluated. Second: external diagnostic cohort, in which diagnostic accuracy of angiography-derived IMR will be assessed in patients with ischemia and no obstructive coronary artery disease (INOCA) and normal controls, whose results were previously published (J Nucl Cardiol. 2020 Sep 30. doi: 10.1007/s12350-020-02252-8.) Among this cohort, 45 patients with no obstructive CAD and normal CZT-SPECT perfusion imaging will be regarded as normal controls, in 35 INOCA patients, vessels with normal corresponding perfusion territory will be regarded as internal control. Third, prognosis cohort, in which 138 consecutive CAD patients received PCI with available angiograms and who were suitable for angiographic fractional flow reserve and IMR measurement will be analyzed. Primary clinical outcome will be cardiac death or congestive heart failure at 2 years from index procedure. Secondary outcome will be any myocardial infarction, ischemia-driven revascularization, definite or probable stent thrombosis, congestive heart failure admission and angina pectoris admission at 2 years from index procedure.

ELIGIBILITY:
Inclusion Criteria:

* CAD patients with available CZT-SPECT within 3 months of measuring FFR in the left anterior descending coronary artery (Cohort 1)
* INOCA patients and normal controls confirmed by CZT-SPECT and angiography (Cohort 2)
* Stable CAD patients received PCI (Cohort 3)
* analyzable angiograms at the index procedure

Exclusion Criteria:

* Previous coronary artery bypass grafting
* Chronic total occlusion patients
* limited image quality of coronary angiography
* Insufficient angiographic project for TIMI frame count
* Severe tortuosity of target vessel
* No optimal projection for reconstruction

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnostic Accuracy Cohort, 53 stable CAD patients who underwent CZT-SPECT MBF and invasive pressure measurements in LAD within 7 days.
  Diagnostic Accuracy Cohort, 35 INOCA patients confirmed by CZT-SPECT and coronary angiography and 45 normal controls Prognosis Cohort 138 stable patients received PCI with available angiograms and who were suitable for angiographic FFR and IMR measurement and have 28 months follow-up data.
Sampling Method: Non-Probability Sample
Enrollment: 271 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | at the index procedure
  Correlation between angiography-derived IMR and HMR
Major adverse cardiac events | at 28 months from index procedure
  Major adverse cardiac events (MACE), including cardiac death and readmission due to heart failure.

SECONDARY OUTCOMES:
A composite of cardiac death, readmission due to heart failure and angina | at 28 months from index procedure
  A composite of cardiac death, readmission due to heart failure and angina
A composite of cardiac death, readmission due to heart failure, spontaneous MI, target vessel revascularization and angina | at 28 months from index procedure
  A composite of cardiac death, readmission due to heart failure, spontaneous MI, target vessel revascularization and angina.
Cardiac death | at 28 months from index procedure
  Cardiac death
Readmission due to heart failure | at 28 months from index procedure
  Readmission due to heart failure
Spontaneous MI | at 28 months from index procedure
  Spontaneous MI
Target vessel revascularization | at 28 months from index procedure
  Target vessel revascularization
Readmission due to angina | at 28 months from index procedure
  Readmission due to angina

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, Professor, Study Chair — Fudan University
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Maria GL, Scarsini R, Shanmuganathan M, Kotronias RA, Terentes-Printzios D, Borlotti A, Langrish JP, Lucking AJ, Choudhury RP, Kharbanda R, Ferreira VM; Oxford Acute Myocardial Infarction (OXAMI) Study Investigators; Channon KM, Garcia-Garcia HM, Banning AP. Angiography-derived index of microcirculatory resistance as a novel, pressure-wire-free tool to assess coronary microcirculation in ST elevation myocardial infarction. Int J Cardiovasc Imaging. 2020 Aug;36(8):1395-1406. doi: 10.1007/s10554-020-01831-7. Epub 2020 May 14. PMID 32409977
- [Result] Ai H, Feng Y, Gong Y, Zheng B, Jin Q, Zhang HP, Sun F, Li J, Chen Y, Huo Y, Huo Y. Coronary Angiography-Derived Index of Microvascular Resistance. Front Physiol. 2020 Dec 16;11:605356. doi: 10.3389/fphys.2020.605356. eCollection 2020. PMID 33391020
- [Derived] Dai N, Che W, Liu L, Zhang W, Yin G, Xu B, Xu Y, Duan S, Yu H, Li C, Yao K, Huang D, Ge J. Diagnostic Value of Angiography-Derived IMR for Coronary Microcirculation and Its Prognostic Implication After PCI. Front Cardiovasc Med. 2021 Oct 15;8:735743. doi: 10.3389/fcvm.2021.735743. eCollection 2021. PMID 34722667